CLINICAL TRIAL: NCT03464422
Title: Adapting an Evidence-based Intervention for Stigma-related Stress, Mental Health, and HIV Risk for MSM of Color in Small Urban Areas (ESTEEM-conneCT)
Brief Title: Adapting an Evidence-based Intervention for Stigma-related Stress, Mental Health, and HIV Risk for MSM of Color in Small Urban Areas
Acronym: ESTEEM-conneCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2000022422; P30MH062294-11 (NIH)
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Results first posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: HIV in MSM
Keywords: HIV; MSM

STUDY DESIGN:
Intervention Model Description: Adaptation of the Effective Skills to Empower Effect Men (ESTEEM; Pachankis, 2014; Pachankis et al, 2015) intervention that addresses young gay and bisexual men's occurring maladaptive behavioral patterns, including HIV-transmission risk behavior and mental health concerns, to address multiple stigma-related stressors for young gay and bisexual men of color in a group therapy format. All participants were part of the same intervention (no randomization) to assess the feasibility and acceptability of this adapted intervention (protocol update 4.24.2019; please see attached protocol). Two cohorts were formed to retain ideal group size for group therapy (10-15 participants per group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Young gay and bisexual men of color (Experimental): Approximately 30 young MSM of color will take part in weekly 90-minute group treatment sessions over 10 weeks. All participants will complete outcome assessments at baseline and three months post-treatment, as well as an exit interview.
  Interventions: Behavioral: ESTEEM conneCT

INTERVENTIONS:
Behavioral: ESTEEM conneCT — The intervention adapts the ESTEEM (Pachankis et al, 2015) intervention to address the multiple-stigma stressors faced by MSM of color, including sexual orientation and racial stigma in a manualized, CBT-based intervention. Approximately thirty participants (divided between two cohorts) will complete ten group sessions will take place at regular times once per week over the course of three months. The groups will be "closed," in that no new members will be allowed to join after the first week in order to promote open self-disclosure and trust among group members.

SUMMARY:
The purpose of this study is adapt an evidence-based intervention for stigma-related stress, mental health, and HIV risk for bay, bisexual, and other men who have sex with men (MSM) of color in small urban areas.

DETAILED DESCRIPTION:
This study has two specific aims. Aim 1 will focus on the modification of an existing intervention manual (created by the study PI) using feedback from previous qualitative interviews with MSM in New Haven and Hartford, CT. Also incorporated will be recent qualitative research on MSM of color's resilience. Specifically, the ways in which racial minority stigma impacts the mental health of MSM in small urban areas and adaptive coping skills that MSM can use in the face of these health threats.

Aim 2, will consist of the deliver of the adapted intervention to approximately 30 young MSM (15 HIV-negative and 15 HIV-positive) to gather data on the feasibility and acceptability of the newly adapted program. The evaluation of the new program will be conducted using pre-post comparisons of quantitative assessments and from qualitative interviews hoped to provide information regarding intervention feasibility, acceptability, and any needed refinement.

This project integrates expertise in culturally-sensitive evidence-based interventions for MSM's HIV risk into a community-based HIV prevention and care context at the Fair Haven Community Health Center, where the intervention will be delivered to the existing patient population.

As of April, 2019, the study protocol was updated and approved by the Yale IRB such that the two intervention cohorts did not differ by HIV serostatus. This decision was made: (1) because of the greater number of HIV-negative men, compared to HIV-positive men, who expressed interest in the study and (2) because participants could decide whether or not to disclose their serostatus in the group, as they do in other real-life interactions with other MSM, as reviewed during the consent process. Thus, there was no group assignment based on HIV serostatus.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

* Report anticipated 6-month residential stability in New Haven county
* Self-identify as a gay or bisexual man or report being a man who has had past-12-month sex with a man
* Self-identify as an ethnic or racial minority, including Black, African American, Caribbean American, Hispanic, and Latinx
* Speak fluent English

Exclusion Criteria:

* Participants not meeting the inclusion criteria will not be eligible to participate.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Identify as men, regardless of sex assigned at birth
Enrollment: 21 (Actual)
Dates: Start 2018-09-09 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Pachankis, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited for the study between September 2018 and February 2019 through local community organizations (e.g., flyers poster at community health clinics, LGBTQ community organizations, university LGBTQ centers) and online (i.e., advertisements posted to Grindr and LGNTQ Facebook groups). Potential participants received a link to a secure online eligibility survey.
Pre-assignment Details: Participants (n = 468) completed an online screener and were contacted for a phone screening (n = 139). Participants who met study inclusion criteria and consented to participate were invited to complete the baseline assessment prior to group assignment (n = 21).
Groups:
- ESTEEM conneCT: ESTEEM conneCT group therapy intervention
Period: Overall Study
Arm/Group | ESTEEM conneCT
Started | 21
Completed | 17
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | ESTEEM ConneCT
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.00 (4.80)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender Identity: Cisgender Man | 20
  Gender Identity: Transgender Man | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Latino/Latinx (Hispanic) | 7
  White (Hispanic) | 5
  Black (Hispanic) | 5
  Black (Non-Hispanic) | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
Sexual Orientation [Count of Participants; unit: Participants]
  Gay | 16
  Bisexual | 3
  Queer | 2
HIV Status [Count of Participants; unit: Participants]
  Negative | 19
  Positive | 2
Income [Count of Participants; unit: Participants]
  Less than $10,000 | 10
  $10,000 - $19,999 | 2
  $20,000 - $29,999 | 2
  $30,000 - $39,999 | 3
  $40,000 - $49,999 | 3
  $50,000 - $74,999 | 1
Education level [Count of Participants; unit: Participants]
  High school diploma or GED | 2
  Some college or Associates degree | 5
  Currently enrolled in college | 2
  4-year college degree (BA, BS, BFA) | 6
  Currently enrolled in graduate school | 3
  Graduate degree | 2
  Some high school | 1

OUTCOME MEASURES:

1. Primary Outcome: Depression
Description: To measure depression in participants, the Center for Epidemiological Studies - Depression Scale (CES-D) will be used. An overall depression score is computed as the sum of the 20 items, with Items 3, 11, 14, and 16 reversed. In cases with internally missing data (items not answered), the sums were computed after imputation of the missing values: # items on scale / # actually answered, multiplied by the sum obtained from the answered items. A higher score indicates more depressive symptomatology during the past week. Range is 0 - 60.
Time Frame: 3 months
Population: Analysis population for 3-month follow-up (n = 17) due to drop out.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM ConneCT
Number analyzed (Participants) | 21
score on a scale
  Baseline | 22.10 (11.89)
  3-month follow-up: number analyzed (Participants) | 17
  3-month follow-up | 20.35 (12.01)

2. Primary Outcome: HIV Transmission Risk
Description: Risk of HIV transmission was assessed through the Past-90-day Timeline Follow-back interview (TLFB; Sobell & Sobell, 1992). HIV risk behavior was calculated as the number of past-90-day sex acts in which key harm-reduction strategies were not employed (e.g., condom, PrEP, viral load suppression) and calculated by dividing the total number of sex acts at risk for HIV transmission by the total number of sex acts. Sex acts range from 0 to (theoretically) infinite.
Time Frame: 90 days
Population: Analysis population for 3-month follow-up (n = 17) due to drop out.
Measure: Mean (Standard Deviation); unit: Number of sex acts conferring HIV risk
Groups:
- ESTEEM ConneCT: ESTEEM ConneCT group therapy
Arm/Group | ESTEEM ConneCT
Number analyzed (Participants) | 21
Number of sex acts conferring HIV risk
  Baseline | 4.10 (10.12)
  3-month follow-up: number analyzed (Participants) | 9
  3-month follow-up | 8.29 (11.38)

3. Secondary Outcome: Overall Depression Severity and Impairment Scale
Description: ODSIS (Bentley et al., 2014) is a 5-item scale that asks individuals to rate the severity and impairment associated with past-week symptoms of depression (e.g., "In the past week, when you have felt depressed, how intense or severe was your depression?) from 0 (little or none: Depression was absent or barely noticeable.) to 4 (extreme: Depression was overwhelming.). Scores range from 0-20, with higher scores indicating greater depression and associated impairment in the past week.
Time Frame: 3 months
Population: Analysis population for 3-month follow-up (n = 17) due to drop out.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM conneCT
Number analyzed (Participants) | 21
score on a scale
  Baseline | 11.00 (4.79)
  3-month follow-up: number analyzed (Participants) | 17
  3-month follow-up | 10.53 (6.07)

4. Secondary Outcome: Overall Anxiety Severity and Impairment Scale
Description: OASIS (Norman et al., 2006) is a 5-item scale that asks individuals to rate the severity and impairment associated with past-week anxiety symptoms (e.g., "In the past week, when you have felt anxious, how intense or severe was your anxiety?") from 0 (little or none: Anxiety was absent or barely noticeable.) to 4 (extreme: Anxiety was overwhelming. It was impossible to relax at all. Physical symptoms were unbearable). Scores range from 0-20, with higher scores indicating greater anxiety and associated impairment in the past week.
Time Frame: 3 months
Population: Analysis population for 3-month follow-up (n = 17) due to drop out.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM ConneCT
Number analyzed (Participants) | 21
score on a scale
  Baseline | 12.05 (3.54)
  3-month follow-up: number analyzed (Participants) | 9
  3-month follow-up | 11.88 (6.07)

5. Secondary Outcome: Brief Symptom Inventory
Description: (BSI; Derogatis & Melisarators, 1983; Meijer et al., 2011). The Global Severity Index of the 18-item BSI provides a mean score across depression, anxiety, and somatization subscales, and assesses psychological distress (e.g., "feeling nervousness or shakiness inside") on a 5-point scale from 0 (not at all) to 4 (extremely) in the past 7 days. Scores range from 0-72, with higher scores indicating worse outcomes (greater symptoms severity).
Time Frame: 3 months
Population: Analysis population for 3-month follow-up (n = 17) due to drop out.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM ConneCT
Number analyzed (Participants) | 21
score on a scale
  Baseline | 2.12 (0.87)
  3-month follow-up: number analyzed (Participants) | 9
  3-month follow-up | 2.05 (1.03)

6. Secondary Outcome: Suicidal Ideation Attributes Scale
Description: SIDAS (van Spijker et al., 2014) is a 5-item scale that assesses past-month frequency and controllability of suicidal thoughts, how close one has come to making an attempt, and distress and impairment associated with thoughts of suicide (e.g., "In the past month, how often have you had thoughts about suicide?"). Responses range from 0 (never or not at all) to 10 (always or extremely) on each item, with item 2 reverse scored. Scale scores range from 0-50, with higher scores indicating more (worse) suicidal ideation
Time Frame: 3 months
Population: Analysis population for 3-month follow-up (n = 17) due to drop out.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM ConneCT
Number analyzed (Participants) | 21
score on a scale
  Baseline | 4.33 (9.63)
  Post-treatment | 3.41 (8.20)

7. Secondary Outcome: Alcohol Use Disorders Identification Test
Description: The AUDIT (Saunders et al.,1993) assesses past-3-month alcohol and related problems across 10 items (e.g., "How often did you have a drink containing alcohol?") with varying numeric response options. A score of 8 or greater serves as a clinical cut-off indicating hazardous drinking. Scores range from 0-40 with higher scores indicating more hazardous drinking (worse outcome)
Time Frame: 3 months
Population: Analysis population for 3-month follow-up (n = 17) due to drop out.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM ConneCT
Number analyzed (Participants) | 21
score on a scale
  Baseline | 16.90 (6.57)
  Post-treatment: number analyzed (Participants) | 9
  Post-treatment | 17.53 (8.77)

8. Secondary Outcome: Condom-use Self-Efficacy Questionnaire
Description: The SSSEQ assesses respondents' confidence in condom use during sex in different scenarios. Example items include, "How confident are you that you could avoid having anal sex without a condom when you are with someone who is really hot?" and "How confident are you that you could avoid having anal sex without a condom when you are drink or high on drugs?". Response options range from 1 (Not at all confident) to 5 (extremely confident). Scores range from 1 - 65 with higher scores indicating greater self-efficacy around practicing safe sex (better outcome)
Time Frame: 3 months
Population: Analysis population for 3-month follow-up (n = 17) due to drop out.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM ConneCT
Number analyzed (Participants) | 12
score on a scale
  Baseline | 48.05 (16.33)
  Post-treatment: number analyzed (Participants) | 9
  Post-treatment | 49.24 (14.32)

9. Secondary Outcome: Sexual Compulsivity Scale
Description: The SCS (Kalichman & Rompa, 2011) assesses respondents' compulsivity around sex. Example items include "My desires to have sex have disrupted my daily life" and "My sexual thoughts and behaviors are causing problems in my life", with response options ranging from 1 (Not at all like me) to 4 (Very much like me). Scores range from 1 - 40 with higher scores indicating greater sexual compulsivity (worse outcome)
Time Frame: 3 months
Population: Analysis population for 3-month follow-up (n = 17) due to drop out.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM ConneCT
Number analyzed (Participants) | 21
score on a scale
  Baseline | 18.38 (7.11)
  3-month follow-up: number analyzed (Participants) | 17
  3-month follow-up | 18.18 (8.89)

10. Secondary Outcome: Gay-Related Rejection Sensitivity Scale
Description: The GRRS (Pachankis, Goldfried & Ramrattan, 2008) asks respondents to rate 14 vignettes in terms of how concerned or anxious each would make them about being rejected because of their sexual orientation, and their likelihood of attributing the rejection to their sexual orientation. For example, one item states, "You've been dating someone for a few years now and you receive a wedding invitation to a straight friend's wedding. The invite was addressed only to you, not you and a guest". Responses to the anxiety and likelihood stems range from 1 (very unconcerned/very unlikely) to 6 (very concerned/very likely). Total score is the sum of the products of anxiety and likelihood scores of all items and ranges from 0-504 with higher scores indicating greater rejection sensitivity (worse outcome).
Time Frame: 3 months
Population: Analysis population for 3-month follow-up (n = 17) due to drop out.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM ConneCT
Number analyzed (Participants) | 21
score on a scale
  Baseline | 10.73 (5.66)
  3-month follow-up: number analyzed (Participants) | 9
  3-month follow-up | 9.92 (5.97)

11. Secondary Outcome: Self-concealment Scale
Description: The SCS (Larson & Chastain, 1990; Schrimshaw, Siegel, Downing & Parsons, 2013) assesses the respondents' concealment of their sexual orientation. Example items include, "I haven't shared with anyone that I have sex with men" and "When I have sex with men, I keep it to myself". Response options range from 1 (strongly disagree) to 5 (strongly agree). Scale scores range from 7-35 with higher scores indicating greater concealment of one's sexual orientation.
Time Frame: 3 months
Population: Analysis population for 3-month follow-up (n = 17) due to drop out.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM ConneCT
Number analyzed (Participants) | 21
score on a scale
  Baseline | 2.15 (0.97)
  3-month follow-up: number analyzed (Participants) | 17
  3-month follow-up | 2.01 (0.95)

12. Secondary Outcome: Internalized Homophobia Scale
Description: The IHS assesses internalized stigma related to respondents' sexual orientation, asking them to rate thoughts and feelings related to their LGBTQ identity (e.g., "You have wished you weren't gay, bisexual, or queer). Responses range from 1 (never) to 4 (often). Scale scores range from 9 - 36 with higher scores indicating greater internalized stigma (worse outcome).
Time Frame: 3 months
Population: Analysis population for 3-month follow-up (n = 17) due to drop out.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM ConneCT
Number analyzed (Participants) | 21
score on a scale
  Baseline | 1.53 (0.68)
  3-month follow-up: number analyzed (Participants) | 17
  3-month follow-up | 1.53 (0.78)

13. Other Pre Specified Outcome: PrEP Use
Description: Participants indicated whether they had been adherent to PrEP in the past three months.
Time Frame: 3 months
Population: Analysis population for 3-month follow-up (n = 17) due to drop out.
Measure: Count of Participants; unit: Participants
Arm/Group | ESTEEM ConneCT
Number analyzed (Participants) | 21
Participants
  Baseline | 6
  3-month follow-up: number analyzed (Participants) | 17
  3-month follow-up | 5

ADVERSE EVENTS:
Time Frame: 3 months
Description: Participants' risk for suicide was assessed at baseline, pre-treatment and post-treatment assessments using the Brief Symptom Inventory (Derogatis & Melisaratos, 1983) and Suicidal Ideation Attributes Scale (Spijker et al, 2014).
Arm/Group | ESTEEM conneCT
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

LIMITATIONS AND CAVEATS:
Protocol was amended (April, 2019) and the cohorts did not differ by HIV serostatus. This decision was made: (1) because of the greater number of HIV-negative men, compared to HIV-positive men, who expressed interest in the study and (2) because participants could decide whether to disclose their serostatus in the group, as they do in other real-life interactions with other MSM, as reviewed during the consent process.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT03464422/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/22/NCT03464422/SAP_001.pdf
  • Informed Consent Form (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT03464422/ICF_002.pdf